CLINICAL TRIAL: NCT06822764
Title: Mental Processes for Rating Pain Intensity
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Erin Dannecker, Assoc Prof, University of Missouri-Columbia
Other Study IDs: 2101603
Record Dates: First submitted 2024-11-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: observational — observational

SUMMARY:
This new study builds on the principal investigator's earlier studies to improve communication about pain. The research team seeks to better understanding of the mental processes needed to rate pain.

ELIGIBILITY:
General inclusion criteria:

* 18 years old or older;
* visited a HCP for treatment of a painful musculoskeletal condition within previous year;
* has usually felt, at least, "mild" musculoskeletal pain on most days of the last 3 months in multiple locations; and
* has felt variable musculoskeletal pain intensity during the last 3 months.

General exclusion criteria:

* past or current employment as a licensed healthcare provider;
* diagnosed with a cardiac arrhythmia;
* has a battery-powered implant in the neck, chest, abdomen, or spine (e.g., pacemaker);
* diagnosed with a neurological condition that causes uncontrolled movement (e.g., Parkinsonism, epilepsy, etc.);
* smokes cigarettes or vapes; (6) has abused substances during the last week; or
* allergic to skin adhesives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 3 weeks
  Pain intensity is the severity or magnitude of perceived pain. The researchers will use a 0 ("no pain")-10("pain as bad as you can imagine") numeric rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States